CLINICAL TRIAL: NCT03459729
Title: PK Analysis of Antitumor B in Patients With Oral Cancer
Brief Title: Pharmacokinetic (PK) Analysis of Antitumor B in Patients With Oral Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stuart Wong, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO36718; R01CA205633 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: Anti-tumor B; ACAPHA; Pharmacokinetics
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Antitumor B; antitumor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antitumor B (Experimental): ATB will be administered on an outpatient basis.
  Interventions: Drug: Antitumor B

INTERVENTIONS:
Drug: Antitumor B — Study participants will take the natural botanical compound ATB during a short window (seven to 28 days). It will be administered at a dose of 1200 mg three times per day (roughly spaced every 8 hours).
  Other Names: Zeng Sheng Ping; ATB; ACAPHA

SUMMARY:
A Window of Opportunity Clinical Trial. This study design permits examination of effects of an oral agent on cancer patients during the "window" between diagnosis of their cancer and their definitive cancer surgery. Similar to a phase 0 study, the trial design permits examination of the biologic effects of an agent; in this study pharmacokinetic properties will be examined.

DETAILED DESCRIPTION:
Study Intervention Description:

Study participants will take the natural botanical compound ATB during a short window (7 to 28 days). Participants will provide blood samples, and saliva samples during Anti-tumor B (ATB) administration and a portion of the initial tumor biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral cavity squamous cell cancer.
* Patient can start study agent administration but histological confirmation of squamous cell cancer (SCC) of the oral cavity (or histologic variants of SCC) by the pathologist must happen within 7 days of registration in order to continue study agent administration.
* Clinical stage II-IVA (as defined by the American Joint Committee on Cancer, 8th Edition [see Amin, 2017]) and amenable to surgical resection
* New diagnosis of oral SCC, new second primary, or recurrent oral SCC following a minimum remission of 6 months following previous definite surgery
* History and physical examination by an otolaryngologist and medical oncologist within 14 calendar days of study registration
* Study agent administration should start within 7 days of registration
* Patient must receive administration of study agent for a minimum of 7 days
* Zubrod Score/Eastern Cooperative Oncology Group (ECOG) Performance status < 2.
* Age ≥ 18 years.
* Complete Blood Count (CBC)/differential obtained within 14 calendar days prior to registration, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3;
  * Platelets ≥ 100,000 cells/mm^3;
  * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.);
* Adequate renal and hepatic function within 14 calendar days prior to registration, defined as follows:

  o Serum creatinine < 1.5 mg/dl or creatinine clearance (CCr) ≥ 50 ml/min within 14 calendar days prior to registration, determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
* Total bilirubin < 2 x the institutional upper limit of normal (ULN) within 14 calendar days prior to registration
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x the institutional ULN within 14 calendar days prior to registration
* Magnesium, calcium, glucose, potassium, and sodium within 14 calendar days prior to registration, with the following required parameters:

  * Magnesium: > 0.9 mg/dl or < 3 mg/dl;
  * Calcium: > 7 mg/dl or < 12.5 mg/dl;
  * Glucose: > 40 mg/dl or < 250 mg/dl;
  * Potassium: > 3 mmol/L or < 6 mmol/L;
  * Sodium: > 130 mmol/L or < 155 mmol/L.
* Female patients must meet one of the following:

  * Postmenopausal for at least one year before the screening visit, or
  * Surgically sterile (e.g., undergone a hysterectomy or bilateral oophorectomy), or
  * If the subject is of childbearing potential (defined as not satisfying either of the above two criteria), agree to practice two acceptable methods of contraception (combination methods requires use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 days after the last dose of study agent, AND
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
* Male patients, even if surgically sterilized (e.g., status post vasectomy), must agree to one of the following:

  * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
  * Must also adhere to the guidelines of any study-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Patients must be deemed able to comply with the study plan.
* Gastric tube study agent administration is permissible.
* Patients must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* History of active liver disease
* Pregnant or lactating women are ineligible due to unforeseeable risks to embryo or fetus.
* Concurrent use of any medicinal botanical, natural, or other herbal compound/s that the study PI believes could potentially impact the results/objectives of this study
* Planned subtotal or debulking surgery, as determined by enrolling physician determination, is not permissible.
* Prior systemic chemotherapy for oral SCC; note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy for oral SCC is permissible if disease free for 1 year since prior oral cancer treatment and free of significant late radiation effects.
* Severe active comorbidity such as uncontrolled cardiac disease, infection, severe Chronic Obstructive Pulmonary Disease (COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six prospective subjects signed the Institutional Review Board-approved consent form. Two subjects did not meet eligibility criteria during screening and were excluded.
Groups:
- Antitumor B: Antitumor B (ATB) will be administered on an outpatient basis.
  Antitumor B: Study participants will take the natural botanical compound ATB during a short window (seven to 28 days). It will be administered at a dose of 1200 mg three times per day (roughly spaced every 8 hours).
Period: Overall Study
Arm/Group | Antitumor B
Started | 6
Received Therapy | 4
Completed | 4
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for Matrine in Saliva
Description: The total systemic exposure to matrine as represented by the AUC will be calculated as the area bounded by the x-axis and the line drawn as straight segments through the plotted matrine concentrations at the time points: predose (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, 360 minutes, 480 minutes, and 1,440 minutes. The results will be reported in (ng x hour)/ml.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng x h/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng x h/mL | 4007.9 (2882.9)

2. Primary Outcome: Area Under the Curve for Matrine in Plasma
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng x h/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng x h/mL | 783.2 (283.7)

3. Primary Outcome: Maximum Concentration (Cmax) of Matrine in Saliva
Description: This measure is the maximum concentration observed. The results will be reported in ng/ml.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng/mL | 457.4 (380.3)

4. Primary Outcome: Maximum Concentration of Matrine in Plasma
Description: This measure is the maximum concentration observed. The results will be reported in ng/ml.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng/mL | 54.5 (14.7)

5. Primary Outcome: Area Under the Curve (AUC) for Maackiain in Saliva
Description: The total systemic exposure to maackiain as represented by the AUC will be calculated as the area bounded by the x-axis and the line drawn as straight segments through the plotted maackiain concentrations at the time points: predose (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, 360 minutes, 480 minutes, and 1,440 minutes. The results will be reported in (ng x hour)/ml.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng x h/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng x h/mL | 0.6 (0.4)

6. Primary Outcome: Area Under the Curve (AUC) for Maackiain in Plasma
Description: as for outcome 5
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng x h/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng x h/mL | 4.4 (3.2)

7. Primary Outcome: Maximum Concentration of Maackiain in Saliva
Description: This measure is the maximum concentration observed. The results will be reported in ng/ml.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng/mL | 0.2 (0.1)

8. Primary Outcome: Maximum Concentration of Maackiain in Plasma
Description: This measure is the maximum concentration observed. The results will be reported in ng/ml.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Antitumor B
Number analyzed (Participants) | 4
ng/mL | 0.3 (0.2)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Antitumor B
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT03459729/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03459729/ICF_001.pdf